CLINICAL TRIAL: NCT05217771
Title: Effect Of High Tone Power Therapy On Selected Symptoms In Post Covid Syndrome
Acronym: WHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Eman Kadry, lecturer assistant, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8976
Record Dates: First submitted 2022-01-24; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High tone power therapy group (Experimental): patients in this group will receive High tone power therapy from 30 to 60 minutes, 3 session /week for 4 weeks with total sessions at least l0 sessions and self-stretch for hand and shoulder.
  Interventions: Other: High tone power therapy group
- control group (Experimental): Patients in control group will receive high tone sham therapy 3 times per week and self-stretch for hand and shoulder.
  Interventions: Other: High tone power therapy group

INTERVENTIONS:
Other: High tone power therapy group — patients in this group will receive High tone power therapy from 30 to 60 minutes, 3 session /week for 4 weeks with total sessions at least l0 sessions and self-stretch for hand and shoulder.

SUMMARY:
The Coronavirus Disease 2019 (COVID-19) is a highly transmittable and pathogenic viral infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2), which emerged in Wuhan, China in December 2019 and its spread around the world has been rapid (Rathi et al., 2021; Vakili et al., 2021). COVID-19 impacts on economy, society, education , neurological, psychiatric and psychosocial impairments , increasing the burden of disease and disability throughout the world have been studied by several authors (Phillips et al., 2020; Pragholapati, 2020).

COVID-19 may lead to greater risks of long-term scarring, permanently lower economic activity, a significant increase in the prevalence of chronic illness, social distancing, isolation, changes in teaching and learning strategies to decrease of number of days of education, the number of social contacts each day is limited (Minister & Majesty, 2020; Almomani et al., 2021) .

DETAILED DESCRIPTION:
The Coronavirus Disease 2019 (COVID-19) is a highly transmittable and pathogenic viral infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2), which emerged in Wuhan, China in December 2019 and its spread around the world has been rapid (Rathi et al., 2021; Vakili et al., 2021). COVID-19 impacts on economy, society, education , neurological, psychiatric and psychosocial impairments , increasing the burden of disease and disability throughout the world have been studied by several authors (Phillips et al., 2020; Pragholapati, 2020).

COVID-19 may lead to greater risks of long-term scarring, permanently lower economic activity, a significant increase in the prevalence of chronic illness, social distancing, isolation, changes in teaching and learning strategies to decrease of number of days of education, the number of social contacts each day is limited (Almomani et al., 2021; Minister & Majesty, 2020) .

Thus, multi-organ injuries are observed in COVID-19, such as acute respiratory distress syndrome, acute myocardial injury, acute kidney injury, and acute liver injury. Survivors of severe COVID-19 are also found to be with multi-organ impairments after discharge (Dennis et al., 2021)

Clinical presentation of COVID- I9 ranges from absence of symptoms to severe pneumonia while fever, dry cough and fatigue, dyspnea, myalgia, arthralgia, distress, anxiety, and depression are common symptoms. The uncommon symptoms include sputum production, headache, hemoptysis, nausea, vomiting and diarrhea among COVID-19 patients (Feng et al., 2020).

Different Phases of COVID-19 defining acute COVID-19 or transition phase: (signs and symptoms of COVID-19 for up to 4 weeks), Acute post COVID symptoms: (signs and symptoms of COVID-19 from 4 to 12 weeks), and long post-COVID-19 syndrome (signs and symptoms that develop during or after an infection consistent with COVID-19, continue for more than 12 weeks up to 24 weeks and are not explained by an alternative diagnosis). persistent post COVID symptoms: symptoms lasting more than 24 weeks (Fernández-de-las-Peñas et al., 2021; Yong, 2021a).

The persisted symptoms of post COVID-19 syndrome are correlated with the severity of illness during acute phase. The illness severity pattern could be categorized as follow; asymptomatic infected patients, symptomatic patients isolating at home, symptomatic patients admitted to hospital, and symptomatic patients requiring ventilatory support in critical care which can lead to permanent sequelae and even death (Castroa et al., 2021).

Persistent post-COVID syndrome (PPCS) or long COVID is a pathologic entity, which involves persistent physical, medical, and cognitive sequelae following COVID-19 as symptoms at least one symptom persists for more than three months after the first symptom onset up to six months. Patients who were no longer positive for SARS-CoV-2 and discharged from the hospital, as well as outpatients, can also develop long COVID (Oronsky et al., 2021).

COVID-19 is a multisystem disease, which in certain cases will require full multidisciplinary team (MDT) rehabilitation required many specialties to enable recovery. The British Society of Rehabilitation Medicine (BSRM) have recently published a position statement that includes the rehabilitation care pathways and coordinated networks that will be required following the COVID-19 pandemic (Barker-Davies et al., 2020).

Rehabilitation may work for treating certain cases of post COVID. There are existing rehabilitation pathways that assess and manage the rehabilitation needs of patients with long-term conditions, notably, cardiac, and pulmonary rehabilitation pathways. These services accommodate patients with multiple comorbidities, including chronic respiratory disease, and cardiovascular, mental health and metabolic diseases. Reviews have also recommended that rehabilitation programs be personalized since post COVID manifestation and pathophysiology may vary in each case (Singh et al., 2020).

High tone power therapy (HiTop) is a new quantum leap in the field of electro therapy without muscle and nerve stimulation. It is electrotherapy with sinusoidal alternating currents. The high tone power therapy provides a therapy with medium frequency sine waves. The therapy is free of direct current (D.C.) components. The amplitude and the frequency are modulated simultaneously. The higher the frequency, the more energy can be introduced corresponding to the individual threshold curve of the patient's electro sensitivity (Medizintechnik, 2008).

High Tone power therapy is increase mitochondria in number and size. The differences in effect relate to two main mechanisms of High Tone power therapy: First, it introduces energy into the body to increase the cell energy potential, to activate cells, to revitalize the body, producing a resonance effect that creates an oscillation or vibration in the cells and tissues. Second, it makes the cell structures oscillate to normalize the metabolism, scattering the mediators of inflammation, nutrients, and waste substances (Requena et al., 2005). so that high tone will be treat persisted symptoms of covid-19.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed with COVID-19 by polymerase chain reaction (PCR) test of a nasopharyngeal sample during acute phase, completed CBC, lymphocyte inflammatory marker, c-reactive protein and ESR.
* Patients must be negative polymerase chain reaction (PCR).
* Patients will be completely recovered from acute symptoms of covid-19.
* Patients will be recruited after 2- 4 weeks post complete recovery from acute symptoms

Exclusion Criteria:

* • Patients with feverish systemic or local bacterial infections.

  * Epilepsy.
  * Pregnant women patients.
  * Cancer.
  * Uncontrolled Diabetes milletus >250 mg/dl

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test | 4 weeks
  for functional capacity
Chalder Fatigue Scale: score can range from 0 to 33, with a higher score indicating greater fatigue. | 4 weeks
  for chronic Fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Emad, Cairo, Egypt